CLINICAL TRIAL: NCT02620150
Title: SSRI Effects on Depression and Immunity in HIV/AIDS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 823405
Record Dates: First submitted 2015-11-20; First posted 2015-12-02 (Estimated); Results first posted 2024-05-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-04

CONDITIONS: Depression; HIV; AIDS
Keywords: HIV; AIDS; Depression; SSRI; Escitalopram; Immunity
MeSH Terms: conditions — Depression; Acquired Immunodeficiency Syndrome | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): CCBT plus Escitalopram, oral, for 10 weeks, once daily, starting at 10mg/day. Tapered up or down, based on tolerability and clinical response, to 20mg/day max.
  Interventions: Drug: Escitalopram
- Placebo (Placebo Comparator): CCBT plus Placebo, oral, for 10 weeks, once daily, starting at 10mg/day. Tapered up or down, based on tolerability and clinical response, to 20mg/day max.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Escitalopram — 10 week trial
  Arms: Experimental
Other: Placebo — 10 week trial
  Arms: Placebo

SUMMARY:
This is a 10 week, double-blind, placebo controlled trial to evaluate SSRI (Selective Serotonin Reuptake Inhibitor) effects for treatment of depression in HIV/AIDS with a focus on innate immunity and inflammation. Depressed population is HIV + on cART (Combination Antiretroviral Therapy), not currently on pharmacotherapy for depression. Subjects will complete computerized cognitive behavior therapy, CCBT for their depression. Blood samples collected for virologic, neuroendocrine, and immunologic evaluation. Our overarching hypothesis is that SSRI treatment of depression and improvement of depressive symptoms leads to increased innate immunity and decreased inflammation, resulting in better control of HIV disease and decreased morbidity.

DETAILED DESCRIPTION:
To pursue our long-term objective of successfully treating co-morbid mental and medical disorders in HIV/AIDS, this study aims to determine whether: 1) SSRI treatment significantly increases innate immunity and decreases chronic inflammation and immune activation, and 2) changes in depressive symptoms correlate with changes in immunity in HIV/AIDS.

HIV-seropositive, depressed subjects will be randomized to 10 weeks of double blind therapy with either escitalopram or placebo. All participants will concurrently begin CCBT (Computerized Cognitive Behavioral Therapy) using the program Good Days Ahead.

Subject visits will occur weekly for the first 6 weeks and then at weeks 8 and 10. The treating clinician will assess side effects, review symptomatic progress, and adjust the study medication as clinically appropriate. An independent clinical evaluator will assess patients at baseline, and weeks 1-6, 8 and 10. Blood samples collected at baseline and weeks 2, 4, and 10 will be used to assay markers of innate immune suppression (lytic units of NK cells, LUNK, and intracellular IFN gamma in NK cells) and markers of inflammation (IL-6 and C-Reactive Protein). At the end of the 10-week treatment phase, all participants will be referred for appropriate clinical treatment of their depression.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 18-70 years, of any race and ethnicity,
2. HIV-seropositive by ELISA and Western Blot assays, infected by behavioral transmission (perinatal HIV excluded),
3. Willing and able to comply with antidepressant medication regimen and scheduled follow-up visits,
4. Currently on a documented regimen of cART for at least 3 months and Viral load less than 200 copies/ml,
5. Current depressive symptoms (HAM-D-17 score ≥ 13 and a SCID diagnosis of either Major Depressive Disorder, Persistent Depressive Disorder (Dysthymia), Unspecified Depressive Disorder, or Other Specified Depressive Disorder)
6. Able to understand and provide informed consent.

Exclusion Criteria:

1. Acute suicidal ideation, gestures, or attempts (e.g., HAM-D suicide item score of 3 "Ideas or gestures of suicide" or 4 "Attempts at suicide" at intake or HAM-D suicide item score of 4 "Attempts at suicide" during study),
2. Significant cognitive impairment or dementia including HIV Associated Dementia (HAD),
3. Use of a medication known to alter immune function within 4 weeks prior to randomization (the following are not excluded: a. acyclovir and related antiviral medications, b. topical corticosteroids, c. corticosteroid nasal sprays or inhalers, d) statin medications,),
4. Immunization with HIV vaccine,
5. Presence of psychotic symptoms or known diagnosis of a primary psychotic disorder,
6. Currently taking an anti-psychotic medication,
7. Pregnant or within nine months post-delivery, lactation,
8. Current or chronic medical condition that would likely preclude adherence to protocol or completion of the trial (per investigator judgment),
9. Bipolar disorder (I or II) or schizophrenia,
10. Current pharmacotherapy for treatment of depression,
11. A history of intolerance or nonresponse to an adequate trial of escitalopram (or other SSRIs),
12. Renal failure, including those who require dialysis,
13. History of epilepsy or seizure disorder,
14. Taken MAOIs within 14 days,
15. On the antibiotic Linezolid and taking IV methylene blue,
16. On a regular regime of medication known to have anticoagulant properties such as NSAID, aspirin or warfarin,
17. A history of acute narrow/closed angle glaucoma,
18. Currently taking CNS drugs (the following are not excluded: gabapentin, pregabalin, varenicline, antihistamines, and hypnotics (e.g. zolpidem, zaleplon, eszopiclone),
19. On any triptan medications,
20. Undergoing ECT.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2017-02-16 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dwight L Evans, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania Perelman School of Medicine, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental | Placebo
Started | 55 | 53
Completed | 48 | 50
Not Completed | 7 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental | Placebo | Total
Number analyzed (Participants) | 55 | 53 | 108
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.95 (11.99) | 49.87 (10.97) | 49.91 (11.45)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 34 | 32 | 66
  Transgender Female | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 7 | 11
  Not Hispanic or Latino | 50 | 46 | 96
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 49 | 47 | 96
  White | 5 | 4 | 9
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 1 | 0 | 1
Overall Score on the Hamilton Depression Rating Scale [Mean (Standard Deviation); unit: units on a scale] — The Hamilton Depression Rating Score (HDRS) score is the sum of 17 items, nine of which takes values 0 through 4 with eight taking values 0 through 2, so the total score ranges from 0 through 52, with higher scores indicating greater severity of depression symptoms. Scores of 0-9 are considered to indicate no/in-remission depression; 10 - 13 mild depression; 14-17 mild to moderate depression; >17 moderate to severe depression.
  units on a scale | 19.13 (4.90) | 19.21 (5.07) | 19.17 (4.96)

OUTCOME MEASURES:

1. Primary Outcome: Natural Killer Cell Activity, Measured in Lytic Units [Bryant J, Day R, Whiteside TL, and Herbeman RB: Calculation of Lytic Units for the Expression of Cell-mediated Cytotoxicity. J Immunol Methods 1992;146:91-103.]
Description: The outcome was determined by biological assays. Natural killer cells (NK cells) are white blood cells, a type of lymphocytes, that destroy infected and cancer cells through antigen independent recognition. Higher numbers indicate higher levels of cytotoxicity, that is, stronger cellular response. In the present summaries, we calculated the within-participant median value of the outcome over their available data at weeks 2, 4 and 10, and obtained overall and within-group summaries for these within-participant distributions.
Time Frame: Post randomization to 10 weeks
Population: 96 participants who provided responses at any of weeks 2, 4, and 10
Measure: Median (Inter-Quartile Range); unit: Lytic Units
Arm/Group | Experimental | Placebo
Number analyzed (Participants) | 46 | 50
Lytic Units | 224.06 [155.81 to 358.33] | 252.02 [150.16 to 360.28]

2. Primary Outcome: Percent of Natural Killer (NK) Cells Producing Intracellular Interferon Gamma (IFN-g)
Description: The outcome was determined by biological assays, which determined the number of NK cells, and the number of these cells that produced IFN-g, and combined these to calculate the outcome. Higher numbers are associated with stronger cellular response. In the present summaries, we calculated the within-participant median value of the outcome over their available data at weeks 2, 4 and 10, and obtained overall and within-group summaries for these within-participant distributions.
Time Frame: Post randomization to 10 weeks
Population: 96 participants who provided responses at any of weeks 2, 4, and 10
Measure: Median (Inter-Quartile Range); unit: Percentage of NK cells producing IFN-g
Arm/Group | Experimental | Placebo
Number analyzed (Participants) | 46 | 50
Percentage of NK cells producing IFN-g | 8.25 [3.50 to 16.00] | 5.40 [3.00 to 11.20]

3. Primary Outcome: Units of Concentration of Plasma Interleukin 6 (IL-6), Expressed as Picograms Per Milliliter
Description: The outcome was determined by biological assays, which determined the concentration of IL-6, expressed as pg/ml. Higher concentrations indicate greater inflammation. In the present summaries, we calculated the within-participant median value of the outcome over their available data at weeks 2, 4 and 10, and obtained overall and within-group summaries for these within-participant distributions.
Time Frame: Post randomization to 10 weeks
Population: 96 participants who provided responses at any of weeks 2, 4, and 10
Measure: Median (Inter-Quartile Range); unit: Concentration of IL-6 (pcg/mL)
Arm/Group | Experimental | Placebo
Number analyzed (Participants) | 46 | 50
Concentration of IL-6 (pcg/mL) | 2.52 [1.57 to 3.71] | 3.17 [2.21 to 4.64]

4. Primary Outcome: Units of Concentration of Plasma C-Reactive Protein (CRP), Expressed as Milligrams Per Liter
Description: The outcome was determined by biological assays, which determined the concentration of CRP, expressed as mg/l. Higher concentrations indicate greater inflammation. In the present summaries, we calculated the within-participant median value of the outcome over their available data at weeks 2, 4 and 10, and obtained overall and within-group summaries for these within-participant distributions.
Time Frame: Post randomization to 10 weeks
Population: 96 participants who provided responses at any of weeks 2, 4, and 10
Measure: Median (Inter-Quartile Range); unit: Concentration of CRP (mg / l)
Arm/Group | Experimental | Placebo
Number analyzed (Participants) | 46 | 50
Concentration of CRP (mg / l) | 3.75 [1.52 to 5.97] | 3.17 [2.21 to 4.64]

5. Secondary Outcome: Correlation Between Change in Overall Score on the Hamilton Depression Rating Scale, and Change in Natural Killer Cell Activity
Description: The outcome was determined by calculating the Spearman correlation between decrease in overall score on the Hamilton Depression Rating Scale and decrease on Natural killer cell activity.
Time Frame: 10 weeks
Population: Participants who provided week 10 Hamilton Depression Rating Scale and Natural Killer cell activity data
Measure: Number; unit: Correlation coefficient
Arm/Group | Experimental | Placebo
Number analyzed (Participants) | 43 | 47
Correlation coefficient | 0.24 | -0.28

6. Secondary Outcome: Correlation Between Change in Overall Score on the Hamilton Depression Rating Scale, and Change in Percent of Natural Killer (NK) Cells Producing Intracellular Interferon Gamma (IFN-g)
Description: The outcome was determined by calculating the Spearman correlation between decrease in overall score on the Hamilton Depression Rating Scale and decrease on the Percent of Natural Killer (NK) Cells Producing Intracellular Interferon Gamma (IFN-g)
Time Frame: 10 weeks
Population: Participants who provided week 10 Hamilton Depression Rating Scale and Intracellular Interferon Gamma (IFN-g) data
Measure: Number; unit: Correlation coefficient
Arm/Group | Experimental | Placebo
Number analyzed (Participants) | 43 | 45
Correlation coefficient | -0.01 | 0.12

7. Secondary Outcome: Correlation Between Change in Overall Score on the Hamilton Depression Rating Scale, and Change in Units of Concentration of Plasma Interleukin 6 (IL-6), Expressed as Picograms Per Milliliter
Description: The outcome was determined by calculating the Spearman correlation between decrease in overall score on the Hamilton Depression Rating Scale and decrease on Units of Concentration of Plasma Interleukin 6 (IL-6)
Time Frame: 10 weeks
Population: Participants who provided week 10 Hamilton Depression Rating Scale and Plasma Interleukin 6 (IL-6) data
Measure: Number; unit: Correlation coefficient
Arm/Group | Experimental | Placebo
Number analyzed (Participants) | 43 | 45
Correlation coefficient | -0.16 | 0.16

8. Secondary Outcome: Correlation Between Change in Overall Score on the Hamilton Depression Rating Scale, and Change in Units of Concentration of Plasma C-Reactive Protein (CRP), Expressed as Milligrams Per Liter
Description: The outcome was determined by calculating the Spearman correlation between decrease in overall score on the Hamilton Depression Rating Scale and decrease on Units of Concentration of Plasma C-Reactive Protein (CRP)
Time Frame: 10 weeks
Population: Participants who provided week 10 Hamilton Depression Rating Scale and Plasma C-Reactive Protein (CRP) data
Measure: Number; unit: Correlation coefficient
Arm/Group | Experimental | Placebo
Number analyzed (Participants) | 43 | 43
Correlation coefficient | -0.33 | -0.04

ADVERSE EVENTS:
Time Frame: 10 weeks
Arm/Group | Experimental | Placebo
All-Cause Mortality (participants affected / at risk) | 1/55 | 0/53
Serious Adverse Events (participants affected / at risk) | 2/55 | 1/53
Other Adverse Events (participants affected / at risk) | 33/55 | 36/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental (N=55) | Placebo (N=53)
Death due to fentanyl/cocaine (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental (N=55) | Placebo (N=53)
Nausea (Gastrointestinal disorders) | 11 | 7
Diarrhea (Gastrointestinal disorders) | 5 | 7
Pain (General disorders) | 6 | 6
Insomnia (Psychiatric disorders) | 4 | 5
Somnolence (Psychiatric disorders) | 4 | 4
Worsening Psychiatric Symptoms (Psychiatric disorders) | 2 | 6
Headache (Nervous system disorders) | 3 | 4
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 | 6
Sexual Dysfunction (General disorders) | 4 | 3
Dry mouth (Nervous system disorders) | 3 | 3
Influenza-like symptoms (General disorders) | 1 | 5
Rash (General disorders) | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-02-09): https://cdn.clinicaltrials.gov/large-docs/50/NCT02620150/Prot_002.pdf
  • Statistical Analysis Plan (2015-03-10): https://cdn.clinicaltrials.gov/large-docs/50/NCT02620150/SAP_001.pdf